CLINICAL TRIAL: NCT05658419
Title: Evaluation of Immediate Loaded Implants Placed Using the Socket Shield Technique in the Esthetic Zone
Brief Title: Immediate Implant vs.Socket Shield Technique in Esthetic Zone
Acronym: Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1103701#
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Bone Loss
Keywords: socket shield
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Study group (socket shield) vs. Control group (immediate implants)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Operator Data collector Examiner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): immediate implant placement
  Interventions: Procedure: socket sheild
- study group (Active Comparator): socket shield immediate implant placement
  Interventions: Procedure: socket sheild

INTERVENTIONS:
Procedure: socket sheild — the socket shield technique, in which a partial root fragment was retained around an immediately placed implant with the aim of avoiding tissue alterations after tooth extraction. Histologic evaluation in a beagle dog showed no resorption of the root fragment and new cementum formed on the implant surface.
  Other Names: partial extraction therapies

SUMMARY:
immediate implant placement versus socket shield approach

DETAILED DESCRIPTION:
This study was a randomized controlled clinical trial; patients were randomly allocated to two groups: the study group: ten dental implants were placed in the maxillary esthetic zone, implants were placed using the socket shield technique with immediate loading; and the control group: ten implants were placed immediately with immediate loading. Preoperative and 6 months postoperative CBCT were performed for both groups to assess the dimensional changes in the labial bone plates. Implant stability quotients (ISQs), pink esthetic scores and attachment loss were measured at the time of implant placement and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patients of 20-45 years of both sexes. Good oral hygiene Demonstrating non-restorable maxillary anterior single rooted teeth in the esthetic zone with as far diagnosable.

Fairly intact buccal periodontal tissues. Patients' acceptance to sign the informed consent. Labial bone plates less than 1.5 mm in thickness or cases with labial root curvatures.

Intact root with no mobility in the tooth and no sub-gingival caries.

Exclusion Criteria:

Patients with systemic diseases that would interfere with the normal healing such as uncontrolled diabetes mellitus.

History of radiation therapy to the head and neck. No history of bruxism/ para-functional habits. (119) Teeth with periodontal disease, vertical root fracture, horizontal fracture at or below the bone level, and teeth with local pathologic incidents that affect the labial part of the root as external or internal root resorption were also excluded.

Maxillary 1st and 2nd premolars. Pregnant and lactating females.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
radiographic bone level | 6 months
  vertical and horizontal bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mohamed Shehata Elsayed, Alexandria, Egypt